CLINICAL TRIAL: NCT00995280
Title: Single Lumen Needle Without Flushing or Double Lumen Needle With Follicle Flushing in Oocyte Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: No sponsor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BHTB-03241705
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Oocyte Retrieval
Keywords: follicle flushing; oocyte retrieval; needle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Single lumen needle use in oocyte retrieval
  Interventions: Device: single lumen needle oocyte retrieval
- 2 (Active Comparator): Double lumen needle with follicle flushing during oocyte retrieval
  Interventions: Device: double lumen needle oocyte retrieval

INTERVENTIONS:
Device: single lumen needle oocyte retrieval — single lumen needle use during oocyte retrieval
  Arms: 1
Device: double lumen needle oocyte retrieval — double lumen needle with 1 time follicle flushing with at least 2 ml during oocyte retrieval
  Arms: 2

SUMMARY:
The aim of this study is to compare whether oocyte flushing during retrieval is effective or not.

DETAILED DESCRIPTION:
In total 300 patients will be randomized for the effectiveness of single or double lumen needle during oocyte retrieval. Double lumen needles give an opportunity of washing to the follicle with flush. Single lumen needles seem to be faster and no need for flushing. We aim to compare to the differences of the use of both needles.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF/ICSI cycles.

Exclusion Criteria:

* Poor responder patients who have lower than 6 follicles at hCG administration day.
* Patients having over 30 follicles.

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Metaphase 2 oocyte number | 6months

SECONDARY OUTCOMES:
clinical pregnancy rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Adana, Turkey (Türkiye)